CLINICAL TRIAL: NCT05128500
Title: Prospective Multicentre Follow-up Evaluating Clinical and Radiological Outcomes of Total Shoulder Arthroplasty With Permedica MIRAI Modular Shoulder Prosthesis System - an Observational Study
Brief Title: Follow-up Evaluating Clinical and Radiological Outcomes of Total Shoulder Arthroplasty With Permedica's MIRAI Prosthesis
Status: Completed | Type: Observational
Sponsor: Permedica spa (Industry)
Responsible Party: Sponsor
Other Study IDs: MIRAI CLH-1
Record Dates: First submitted 2021-11-09; First posted 2021-11-22 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Cuff Tear Arthropathy; Primary Osteoarthritis; Secondary Osteoarthritis; Shoulder Osteoarthritis; Rheumatoid Arthritis Shoulder; Psoriatic Arthritis; Fracture, Shoulder; Avascular Necrosis of Humerus
Keywords: Total Shoulder Arthroplasty; Shoulder Prosthesis; Observational Study; Cuff Tear Arthropathy; Shoulder Osteoarthritis
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy; Arthritis, Psoriatic; Shoulder Fractures | interventions — Arthroplasty, Replacement, Shoulder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Total Shoulder Arthroplasty with Permedica's MIRAI — Total Shoulder Arthroplasty with Permedica's MIRAI Modular Shoulder Prosthesis System

SUMMARY:
This observational study is conducted in order to evaluate the effectiveness of the primary total shoulder arthroplasty with the Permedica's MIRAI Modular Shoulder Prosthesis System on the general population of patients who are about to undergo this surgery for every indication. Patients requiring a revision shoulder arthroplasty will not be enrolled.

The effectiveness will be evaluated in terms of recovery of shoulder function and stability of the prosthetic implant. The incidence of complications, adverse and serious adverse events will also be studied. Additional study aim is to evaluate a medium/long term survival of the prosthesis.

The duration of the study per single subject is 5 years.

ELIGIBILITY:
Inclusion Criteria:

* both genders
* at least 18 years old of age
* undergoing a primary total shoulder arthroplasty with MIRAI® Prosthesis System (anatomic or reverse, stemless or stemmed).
* Signed informed consent

Exclusion Criteria:

* Patients requiring a revision shoulder arthroplasty
* Persistent chronic or acute infections and all septic conditions
* Persistent osteomyelitis local or systemic
* Allergy or hypersensitivity to the substances contained in the materials of the implanted components
* Acute or chronic neurological and/or musculoskeletal impairment which compromises the shoulder joint function such as an axillary nerve injury affecting the deltoid muscle
* Inadequate bone structure which cannot guarantee stability to the prosthetic components
* Several vascular, nerve or muscular disorders, which compromise related extremities
* Marked osteoporosis, osteomalacia
* Hypotrophy of the periarticular soft tissues
* Dysmetabolic diseases such as, for example, kidney failure or systemic diseases
* Muscular insufficiency
* Active neoplastic or metastatic diseases
* Any other clinical or physical condition that can invalidate the surgery, the rehabilitation or the prosthesis stability
* Patient unwilling or unable to undergo the rehabilitation or to return to follow-up visits
* Women in pregnancy, childbearing potential or breastfeeding
* Involvement in other ongoing studies or clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are about to undergo a primary total shoulder arthroplasty in daily clinical practice, referring to one of the project investigator at the study site will be proposed to partecipate to the study.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Clinical outcome: Change of shoulder function | 5 years
  Change of "American Shoulder and Elbow Surgeons" (ASES) Score. Total score 0-100 ASES points, 0 = worse pain and functional loss/disability.
Clinical outcome: Change of shoulder function | 5 years
  Change of "Disabilities of the Arm, Shoulder and Hand" (DASH) Score. A higher score indicates greater disability. DASH disability/symptom score = [(sum of n responses) - 1]/n x 25, where n is equal to the number of completed responses.
Clinical outcome: Change of shoulder function | 5 years
  Change of Constant Score. Total score 0-100 Constant points, 0 = worse outcome and functional loss/disability; 100 = better outcome, shoulder function improvement.
Clinical outcome: Change of shoulder function | 5 years
  Change of active Range of Motion (ROM)

SECONDARY OUTCOMES:
Radiological outcome: Radiological implant stability | 5 years
  Presence of Radiolucent Lines and other radiological signs of instability
Radiological outcome: Radiological implant stability | 2 years
  Presence of Radiolucent Lines and other radiological signs of instability
Safety Outcome | 5 years
  Incidence of adverse events and complications
Implant survival rate | 5 years
  Rate of revisions. Survival estimated with Kaplan-Meier method.
Implant survival rate | 2 years
  Implant failures. Survival estimated with Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Banci, Study Director — Permedica
Locations (4):
- Germany (2):
  - go:h - Gelenkchirurgie Orthopädie: Hannover, Hanover
  - Krankenhaus Reinbek St. Adolf-Stilt, Reinbek
- ULSS 1 Dolomiti - Presidio Ospedaliero Santa Maria del Prato di Feltre, Feltre, Italy
- Orthopädische Klinik Luzern - OKL, Lucerne, Switzerland